CLINICAL TRIAL: NCT04052711
Title: A Randomized, Controlled Study to Evaluate the Sensitizing Potential of FMX-101 in Healthy Volunteers Using a Repeat Insult Patch Test Design
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FX2016-07
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Healthy
MeSH Terms: interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FMX-101 (Experimental)
  Interventions: Drug: FMX-101

INTERVENTIONS:
Drug: FMX-101

SUMMARY:
A Randomized, Controlled Study to Evaluate the Sensitizing Potential of FMX-101 in Healthy Volunteers Using a Repeat Insult Patch Test Design

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 and older who was healthy
2. Was of any Fitzpatrick Skin Type or race, providing the skin pigmentation allowed for discernment of erythema

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2016-11-19 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
Assessment of recurrence of a cutaneous response at Rechallenge equivalent to or more severe than that observed at Challenge. | 8 weeks